CLINICAL TRIAL: NCT07355777
Title: Prospective Multicenter Randomized Trial Comparing Oral Explanation Alone and With Video Tutorial for Bowel Preparation Quality and Adenoma Detection
Brief Title: Video Tutorial and Oral Explanation Vs Oral Explanation Alone in Colonoscopy Preparation
Acronym: PREPACOTUTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Collaborators: Clinique Charcot (Unknown); Clinique du Val d'ouest (Unknown); Infirmerie Protestante de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PREPACO -TUTO
Record Dates: First submitted 2025-09-29; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Colonoscopy; Gastro-Intestinal Disorder
Keywords: colon preparation; colonoscopy; gastro-intestinal disorder; tutorial
MeSH Terms: conditions — Digestive System Diseases | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- face to face + Tutorial (Experimental): one arm F+T "face to face + Tutorial" will have, in addition to all the items received by Group F, an email containing a link to a video tutorial explaining how to perform colonic preparation.
  Interventions: Procedure: Colonoscopy
- face to face (Active Comparator): The other arm F : "face to face" of patients will have the explanation of the colonic preparation and the administrative and legal documents of the centre's current practice by the gastro-enterologist.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — The explanation of the colonic preparation will be done at home by film tutorial, before the colonic procedure or as usual, by the physician during a specific consultation before the colonic procedure but the quality of preparation will be evaluated by the boston score as usual.

SUMMARY:
Colonoscopy which is the standard examination for the exploration of the colon and rectum is performed very frequently.

Colon preparation before the examination is an essential step and pescription of the colonic preparation is carried out by the gastroenterologist.

However, despite a standardized explanation of the colon preparation, there is heterogeneity in understanding the colonic preparation, which in some cases compromises the quality of the colonoscopy examination. This clinical study aims to investigate whether an explanation of colonic preparation by tutorial films would increase the quality of colon preparation and would reach the recommendations of the Société française d'endoscopie digestive (SFED) in 2019.

DETAILED DESCRIPTION:
The quality of the colonic preparation is essential for the quality of the colonic examination: in one hand, a good preparation will allow the feasibility of the colonoscopy and will allow a complete examination. On the other hand, the presence of stercoral residues due to a bad colonic preparation reduces the sensitivity of the examination by hiding small lesions or with a very discreet relief. A poorer quality will also increase the length of the examination, which increase the risk of complications. However, in the literature, 20 to 30% of poor colonic preparation is found and 5% of colonoscopies are incomplete, including 42% due to poor preparation. The Pacôme survey, reveals that 6% of patients did not have prior consultation with the gastroenterologist. In addition, if 81% of patients were informed of the importance of the preparation, only 64% were aware of its practical modalities. Only 57% of patients were aware of the risks of inadequate preparation, despite the fact that doctors feel they have well informed their patients. It is also reported in "2 days of endoscopy 2008", that 8% of the information is given by someone other than the gastroenterologist himself. These data demonstrate that there is a heterogeneity in the explanatory content of the consultation prior to the colonoscopy examination. This can then explain the rate of poor quality colonic preparation and consequently the colonoscopy examination. The consultation must be a real therapeutic education and must be sufficiently informative to result in a colonic preparation of quality. We then hypothesize that an informative explanation in the form of a tutorial film would ensure homogeneous and standardized information between practitioners. In addition, the tutorial film will be available to be viewed at home several times by the patient, which may reduce the risk of misunderstanding.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing their first colonoscopy for gastrointestinal symptoms, family history of CRC or suspected CRC.
* Ability to use the internet and a link to a video.
* Life expectancy over three months.
* Patient ≥ 18 years old, requiring a colonoscopy procedure.

Exclusion Criteria:

* Patient with any psychiatric or psychological disorder that does not allow them a properd understanding and follow-up of the study.
* Patient without internet access.
* Patient requiring a colonoscopy procedure in emergency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the quality of the colonic preparation by the boston score for each groupe | During the colonoscopy procedure
  To date, the evaluation of the quality of the colonic preparation recognized by the SFED is the establishment of the Boston score. For each group, calculate the percentage of patients obtaining a Boston score ≥ 7.
  A Boston score ≥ 7 for a high-quality preparation is the score to be obtained according to the 2019 SFED recommendations for at least 90% of patients, excluding colonoscopies performed for emergencies.

SECONDARY OUTCOMES:
Detection rate of adenomas in each arm will be compared | During the colonoscopy procedure
  Number of patients with the detection rate of adenomas in each group will be compared in order to determine if there is a difference of sensibility between the two types of colonic explanation
The rate of complete colonoscopy in each group | During the colonoscopy procedure
  Number of patients with complete colonoscopy in each group will be compared in order to determine if there is a difference of faisability between the two types of colonic explanation.
Incidence of procedure- adverse events as assessed by complications reports | From the colonoscopy procedure to one day after
  Number of patients with procedure-related adverse events will be reported to the pharmacovigilance department.

CONTACTS AND LOCATIONS:
Overall Officials: Marc O'BRIEN, Principal Investigator — Hopital Saint Joseph Saint Luc
Locations (5):
- France (5):
  - Saint Joseph Saint Luc Hospital, Lyon, RHONE-ALPES, Lyon
  - Clinique De L'infirmerie Protestante 3 Chem. du Penthod 69300 Caluire-et-Cuire, Lyon
  - Clinique du Val d'ouest 39 chemin de la Vernique 69130 Ecully, Lyon
  - Clinique Médico-Chirurgicale Charcot 51 rue Commandant Charcot 69110 Sainte-Foy-lès-lyon, Lyon
  - Les portes du sud 2 avenue du 11 novembre 1918 69200 Vénissieux, Lyon